CLINICAL TRIAL: NCT02169765
Title: Hepatic Resection Versus Radiofrequency Ablation for Early-stage Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: HR Versus RFA for Early Stage HCC
Acronym: ARTC-HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Affiliated Tumor Hospital, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRRFA-HCC; HRRFA-HCC (Registry Identifier: Jian-Hong Zhong)
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatic resection (Active Comparator): Indications for HR were the presence of appropriate residual liver volume determined by volumetric computed tomography and lack of hepatic encephalopathy.
  Interventions: Other: Hepatic resection
- Radiofrequency ablation (Experimental): Radiofrequency ablation is performed in less than one week after clinical diagnosis.
  Interventions: Other: Radiofrequency ablation

INTERVENTIONS:
Other: Hepatic resection — Adequate remnant liver volume was 30% for HCC patients without cirrhosis, and >50% for HCC patients with chronic hepatitis, cirrhosis, or severe fatty liver.
  Arms: Hepatic resection
Other: Radiofrequency ablation — Radiofrequency ablation is performed in less than one week after clinical diagnosis.
  Arms: Radiofrequency ablation

SUMMARY:
Hepatocellular carcinoma (HCC) is the third leading death cancer in the world. It is important to explore a safe and effective therapy for early-stage HCC. Previous studies reported that radiofrequency ablation (RFA) has higher efficacy and is associated with fewer complications and shorter hospital stays than hepatic resection (HR) for early-stage HCC. However, meta-analysis and systematic review found that RFA is associated with higher recurrence rate and lower long-term overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Clinical diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients
* Tumor stage fitted into Milan Criteria
* Patients have Child-Pugh A liver function
* No previous neoadjuvant treatment
* No evidence of metastasis to the lymph nodes and/or distant metastases on the basis of preoperative imaging results and perioperative findings
* No malignancy other than HCC for 5 years prior to the initial HCC treatment
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding

Exclusion Criteria:

* History of cardiac disease:

  * Congestive heart failure > New York Heart Association (NYHA) class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted);
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; or
  * Uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections ( > grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survivals | 5-years

SECONDARY OUTCOMES:
Recurrence rates | 5-years

OTHER OUTCOMES:
morbidity | 30,90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

REFERENCES:
- [Background] Cho YK, Rhim H, Noh S. Radiofrequency ablation versus surgical resection as primary treatment of hepatocellular carcinoma meeting the Milan criteria: a systematic review. J Gastroenterol Hepatol. 2011 Sep;26(9):1354-60. doi: 10.1111/j.1440-1746.2011.06812.x. PMID 21679247
- [Background] Cucchetti A, Piscaglia F, Cescon M, Colecchia A, Ercolani G, Bolondi L, Pinna AD. Cost-effectiveness of hepatic resection versus percutaneous radiofrequency ablation for early hepatocellular carcinoma. J Hepatol. 2013 Aug;59(2):300-7. doi: 10.1016/j.jhep.2013.04.009. Epub 2013 Apr 18. PMID 23603669
- [Background] Duan C, Liu M, Zhang Z, Ma K, Bie P. Radiofrequency ablation versus hepatic resection for the treatment of early-stage hepatocellular carcinoma meeting Milan criteria: a systematic review and meta-analysis. World J Surg Oncol. 2013 Aug 13;11(1):190. doi: 10.1186/1477-7819-11-190. PMID 23941614
- [Background] Wang Y, Luo Q, Li Y, Deng S, Wei S, Li X. Radiofrequency ablation versus hepatic resection for small hepatocellular carcinomas: a meta-analysis of randomized and nonrandomized controlled trials. PLoS One. 2014 Jan 3;9(1):e84484. doi: 10.1371/journal.pone.0084484. eCollection 2014. PMID 24404166
- [Background] Cho YK, Kim JK, Kim WT, Chung JW. Hepatic resection versus radiofrequency ablation for very early stage hepatocellular carcinoma: a Markov model analysis. Hepatology. 2010 Apr;51(4):1284-90. doi: 10.1002/hep.23466. PMID 20099299